CLINICAL TRIAL: NCT00342927
Title: Family Investigation of Nephropathy and Diabetes (F.I.N.D.)
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999901117; 01-DK-N117
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-06-03

CONDITIONS: Diabetic Nephropathy; Diabetes Mellitus; Diabetic Kidney Disease; Albuminuria
Keywords: American Indians; Complications; Genetics; Linkage; Type 2 Diabetes; Natural History; Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus; Albuminuria; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Volunteers: Volunteers for a genetic study of diabetes and nephropathy

SUMMARY:
The Family Investigation of Nephropathy and Diabetes (FIND) is a multicenter study designed to identify genetic determinants of diabetic kidney disease. FIND will be conducted in eleven centers and in many ethnic groups throughout the United States. Two different strategies will be used to localize genes predisposing to kidney disease: a family-based genetic linkage study and a case-control study that utilizes admixture linkage disequilibrium. The center based at the Phoenix office of the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK-Phoenix) will conduct family-based linkage studies among American Indian populations in the southwestern United States.

Participants (index cases) with diabetes and kidney disease will initially be recruited, and their parents and siblings will also be invited to participate. Genetic material from these participants will be used to genotype markers throughout the genome. Linkage analysis will be conducted to identify particular chromosomal regions containing genes that influence susceptibility to diabetic kidney disease. Linkage analyses will also be used to identify genes influencing traits related to diabetic kidney disease, such as serum creatinine, urinary protein excretion, plasma glucose levels, blood pressure and blood lipid levels. Regions that show evidence for linkage will then be examined in more detail, with both genetic linkage and association studies, to attempt to identify the specific genes that influence diabetic kidney disease, or related traits.

The identification of genes that influence susceptibility to diabetic kidney disease will lead to a better understanding of how kidney disease develops. In the long run, this may lead to improved treatment and prevention of diabetic kidney disease....

DETAILED DESCRIPTION:
The Family Investigation of Nephropathy and Diabetes (FIND) is a multicenter study designed to identify genetic determinants of diabetic kidney disease. FIND is conducted in eleven centers and in many ethnic groups throughout the United States. Two different strategies are used to localize genes predisposing to kidney disease: a family-based genetic linkage/association study and a case-control study that uses admixture linkage disequilibrium. The center based at the Phoenix office of the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK-Phoenix) conducts family-based linkage/association studies among American Indian populations in the southwestern United States, and in the indigenous Micronesian populations of the Territory of Guam and the Commonwealth of the Northern Mariana Islands (CNMI).

Participants (index cases) with diabetes and kidney disease are recruited, and their parents and siblings are also invited to participate. Members of target populations who are not related to index cases are also included and offered screening for diabetes and kidney disease; this will facilitate association studies. Genetic material from these participants is used to genotype markers throughout the genome. Linkage and association analyses are conducted to identify particular chromosomal regions containing genes that influence susceptibility to diabetic kidney disease. Linkage and association analyses are also used to identify genes influencing traits related to diabetic kidney disease, such as serum creatinine, urinary protein excretion, plasma glucose levels, blood pressure and blood lipid levels. Genome-wide and candidate gene association studies are also conducted. Regions that show evidence for linkage or association are then examined in more detail, with both genetic linkage and association studies, to attempt to identify the specific genes that influence diabetic kidney disease, or related traits.

The identification of genes that influence susceptibility to diabetic kidney disease will lead to a better understanding of how kidney disease develops. In the long run, this may lead to improved treatment and prevention of diabetic kidney disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

Index Cases:

Individuals with diabetes and diabetic nephropathy who are at least 18 years of age.

Potential index cases must have at least one sibling, or both parents available as potential study participants.

Potential index cases must also have diabetic nephropathy. An index case must have nephropathy that is more severe than microalbuminuria. An index case must meet one of the following criteria:

1. Biopsy proven diabetic nephropathy (by medical record review):

   1. Nodular and/or diffuse increases in the mesangial matrix accumulation; and
   2. Thickened glomerular basement membranes and/or arteriolar hyalinization; and
   3. Absence of mesangial immunoglobulin or paraprotein deposits by immunoflorecscence microscopy, absence of amyloid deposits by Congo Red staining or electron microscopy, absence of electron dense deposits within the glomerular basement membrane or glomerular capillary subendothelial space; and
   4. Overt proteinuria, defined as ACR greater than or equal to 300 mg/g, urinary protein creatinine ratio greater than or equal to 0.5 g/g, urinary albumin excretion greater than or equal to 300 mg/24 hr, or urinary protein excretion greater than or equal to 0.5 g/24 hr.
2. ESRD (including transplant) from presumed diabetic nephropathy:

   Diabetes present for at least 5 years prior to the initiation of replacement therapy and retinopathy at any time;

   or Diabetes present for at least 5 years prior to the initiation of replacement therapy and either greater than or equal to 3 gm protein/24 hours, or a urine protein (mg)/creatinine (mg) greater than or equal to 3.0 or urinary ACR greater than or equal to 3000 mg/g or urinary albumin excretion greater than or equal to 3000 mg/24 hours (historical data acceptable);

   or retinopathy and either greater than or equal to 3 gm protein/24 hours, or a urine protein (mg)/creatinine (mg) greater than 3.0 or urinary ACR greater than or equal to 3000 mg/g or urinary albumin excretion greater than 3000 mg/24 hours (historical data acceptable).
3. Patient with presumed diabetic nephropathy but not ESRD:

Patient has diabetic retinopathy and either greater than or equal to 1 gram proteinuria/24 hours or a urine protein (mg)/creatinine (mg) greater than or equal to 1.0 or urinary ACR greater than or equal to 1000 mg/g or urinary albumin excretion greater than or equal to 1000 mg/24 hours (historical data acceptable);

or first detection of either greater than or equal to 3 gram protein/24 hours or a urine protein (mg)/creatinine (mg) greater than or equal to 3.0 gram or urinary ACR greater than or equal to 3000 mg/g or urinary albumin excretion greater than or equal to 3000 mg/24 hours at DM duration greater than or equal to 10 years (historical data acceptable).

Recruitment of Family Members:

Any available parent or sibling who is at least 18 years of age will be recruited as a potential participant and will use the same criteria as above.

DNA for individuals in informative families will be submitted to the genotyping laboratory. An informative family is defined as one for which DNA specimens are available for the following individuals:

1. The index case and both parents, or
2. The index case and at least one other affected sibling who has diabetes and renal disease, or
3. The index case and at least one unaffected sibling, defined as an individual who has had diabetes for at least 10 years and who has no renal disease (based on evidence obtained from the medical record and from the FIND examination.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers from the community
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2001-03-07 (Actual)

PRIMARY OUTCOMES:
Diabetes and diabetic kidney disease. | throughout the study
  Diabetes and kidney disease ascertained through diagnostic tests.

SECONDARY OUTCOMES:
Blood pressure and serum lipids. | throughout the study
  Blood pressure measurement and serum lipids by laboratory analysis

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Hanson, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided